CLINICAL TRIAL: NCT05349695
Title: Patient Profiling and Outcome Assessment in Spinal Cord Stimulation for Chronic Back and/or Leg Pain: Study Protocol for a Prospective, Multicentric Observational Study (the PROSTIM Study)
Brief Title: Patient Profiling and Outcome Assessment in Spinal Cord Stimulation for Chronic Back and/or Leg Pain
Acronym: PROSTIM
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Studie- & Opleidingscentrum Neurochirurgie Virga Jesse (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Principal Investigator, Mark Plazier, Prof. Dr. Plazier, Studie- & Opleidingscentrum Neurochirurgie Virga Jesse
Other Study IDs: 001
Record Dates: First submitted 2022-04-12; First posted 2022-04-27 (Actual); Last update posted 2022-04-27 (Actual); Status verified 2022-04

CONDITIONS: Failed Back Surgery Syndrome; Chronic Pain
Keywords: Spinal cord stimulation; Patient profiling; Treatment pathways; Outcome assessment; Medial pathway; Lateral pathway; Descending pain modulation
MeSH Terms: conditions — Failed Back Surgery Syndrome; Chronic Pain | interventions — Spinal Cord Stimulation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Spinal cord stimulation — Eligible patients will undergo a SCS trial period for three weeks (as legally defined by the reimbursement authorities). The leads can be placed both surgically of percutaneously with an external trial stimulator. Surgical implantation of an implanted pulse generator (IPG) is performed if the patient achieves at least 50% pain reduction and a reduced pain medication use (reimbursement requirements) during the trial period. Subsequently, the implanted devices are programmed to the optimal parameters in collaboration with a nurse specialized in SCS treatment. The patients are educated on the use of the patient programmer.

SUMMARY:
The PROSTIM study is an ongoing prospective, multicentric and observational clinical study. Patients are recruited in three different centers in Eastern Belgium from May 2018 onwards. This real-world data collection approaches the outcome assessment of daily medical practice. A hierarchical cluster analysis is used to identify significant patient clusters based on the Visual Analogue Scale (VAS), Oswestry disability index (ODI), Pain Vigilance and Awareness Questionnaire (PVAQ), Pain Catastrophizing Scale (PCS) and EuroQol with five dimensions for health-related quality of life (EQ-5D). Patient clusters will be assessed on the change in biopsychosocial variables after six weeks, three and twelve months. Secondary outcomes include the comparison of pain medication use, SCS parameters, treatment satisfaction and return to work.

ELIGIBILITY:
Inclusion Criteria:

* Male/female over 18 years old.
* Chronic intractable back and/or leg pain (PSPS T2), refractory to conservative treatment measures.
* Positive recommendation after multidisciplinary assessment including psychiatric assessment.
* Patients are capable of giving written informed consent.

Exclusion Criteria:

* Negative recommendation after multidisciplinary assessment (ex. psychiatric disorders).
* Insufficient improvement during trial period.
* Previous SCS implantation.
* Removal due to complication (infection, loss of function,...)
* Surgical contraindication (infection of surgical site, coagulation disorders,..)
* Pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of patients with chronic back and/or leg pain who have been approved by the multidisciplinary team for SCS treatment.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-05-01 (Estimated); Primary Completion 2023-05 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
Back pain | 3 weeks
  Visual analogue scale back (0-10)
Leg pain | 3 weeks
  Visual analogue scale back (0-10)
Back pain | 6 months
  Visual analogue scale back (0-10)
Leg pain | 6 months
  Visual analogue scale back (0-10)
Back pain | 12 months
  Visual analogue scale back (0-10)
Leg pain | 12 months
  Visual analogue scale back (0-10)
Disability | 3 weeks
  Oswestry Disability Index, ODI (0-100)
Disability | 6 months
  Oswestry Disability Index, ODI (0-100)
Disability | 12 months
  Oswestry Disability Index, ODI (0-100)
Health-related quality of life | 3 weeks
  EQ-5D-3L
Health-related quality of life | 6 months
  EQ-5D-3L
Health-related quality of life | 12 months
  EQ-5D-3L

SECONDARY OUTCOMES:
Pain medication | 3 weeks
  WHO classification and/or the use of neuropathic pain medication
Pain medication | 6 months
  WHO classification and/or the use of neuropathic pain medication
Pain medication | 12 months
  WHO classification and/or the use of neuropathic pain medication
Spinal cord stimulation type | 3 weeks
  Type of spinal cord stimulation amongst different patient clusters
Spinal cord stimulation type | 6 months
  Type of spinal cord stimulation amongst different patient clusters
Spinal cord stimulation type | 12 months
  Type of spinal cord stimulation amongst different patient clusters
Satisfied with current treatment | 3 weeks
  Yes/No question
Satisfied with current treatment | 6 months
  Yes/No question
Satisfied with current treatment | 12 months
  Yes/No question
Rate of return to work | 3 weeks
  % of patients returning to work or daily activities
Rate of return to work | 6 months
  % of patients returning to work or daily activities
Rate of return to work | 12 months
  % of patients returning to work or daily activities

CONTACTS AND LOCATIONS:
Overall Officials: Mark Plazier, MD,PhD, Principal Investigator — Jessa Hospital Hasselt, Belgium
Locations (3):
- Belgium (3):
  - Jessa Hospital, Hasselt
  - Sint-Franciscus Ziekenhuis, Heusden-Zolder
  - St. Trudo Ziekenhuis, Sint-Truiden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Raymaekers V, Meeuws S, Goudman L, der Steen GV, Moens M, Vanloon M, Ridder D, Menovsky T, Vesper J, Plazier M. Patient profiling and outcome assessment in spinal cord stimulation for chronic back and/or leg pain (the PROSTIM study): a study protocol. Pain Manag. 2023 Dec;13(12):677-687. doi: 10.2217/pmt-2023-0103. Epub 2023 Dec 6. PMID 38054386